CLINICAL TRIAL: NCT02894684
Title: Aztreonam for Inhalation Solution (AZLI) for the Treatment of Exacerbations of Cystic Fibrosis. An Randomised, Crossover Pilot Study of AZLI Plus Intravenous Colistin® Versus Standard Dual Intravenous Therapy
Brief Title: Aztreonam for Inhalation Solution (AZLI) for the Treatment of Exacerbations of Cystic Fibrosis
Acronym: AZTEC-CF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016AZLIND001
Record Dates: First submitted 2016-09-01; First posted 2016-09-09 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Cystic Fibrosis; Infection; Pseudomonas
MeSH Terms: conditions — Cystic Fibrosis; Infections; Pseudomonas Infections | interventions — Aztreonam; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZLI then Standard Care (Experimental): Upon first exacerbation this arm will receive AZLI, on their second they will receive standard care
  Interventions: Drug: Aztreonam; Drug: Standard Care
- Standard Care then AZLI (Active Comparator): Upon first exacerbation this arm will receive standard care, on the second exacerbation this arm will receive AZLI
  Interventions: Drug: Aztreonam; Drug: Standard Care

INTERVENTIONS:
Drug: Aztreonam — 14 days of AZLI: 75mg TDS PLUS IV Colistin
  Other Names: Cayston; AZLI
Drug: Standard Care — 14 days of IV Colistin plus one of Tazocin/Ceftazidime/Meropenem/Aztreonam/Fosfomycin

SUMMARY:
This study evaluates the role of AZLI in the treatment of acute pulmonary exacerbations of CF. For consecutive exacerbations patients will receive AZLI + IV Colistin, or two IV anti-pseudomonals.

DETAILED DESCRIPTION:
AZLI, marketed as Cayston, is an inhaled beta-lactam antibiotic. It has a license for the chronic suppression of Pseudomonas aeruginosa (PA). Current standard practice dictates the use of two IV antipseudomonal antibiotics for the treatment of acute pulmonary exacerbations. The increasing survival, and hence population, in CF means that newer antimicrobial strategies are required in order to manage antimicrobial resistance, minimise adverse systemic effects of heavy antimicrobial exposure and also make effective use of resources. Inhaled antibiotics are commonly used in the chronic suppression of PA yet their use has not been thoroughly investigated in acute pulmonary exacerbation. Inhaled antibiotics deliver their drugs directly to the target-site with minimal systemic absorbance, making them an attractive candidate for treatment of acute exacerbations.

Recently, it has become apparent that the bacterial community is much more complex than initially thought. The microbiome, a term used to describe the polymicrobial community in the lungs, has become apparent due to the use of modern culture-independent methods to detect bacteria. The microbiome changes in composition and structure around the time of exacerbations and in response to treatment, although these changes have not been prospectively characterised.

We have designed an open-label randomised, controlled cross-over trial to investigate the clinical effectiveness of of AZLI in the treatment of acute pulmonary exacerbation, whilst simultaneously comparing the effect inhaled and intravenous antibiotics have on the microbiome.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of CF
2. Patients aged 18 - 65 years of age who can give informed consent
3. FEV1 >25% or <75% predicted (in keeping with Cayston® license)
4. Admitted to the Liverpool Heart & Chest Hospital with an exacerbation of CF pulmonary disease
5. Presence of PA in lower respiratory tract cultures in the 6 months prior

Exclusion Criteria:

1. Documented allergy to beta-lactam antibiotics or IV Colistin
2. Growth of Burkholderia Cepacia Complex (BCC) within 2 years
3. Pregnancy
4. Previous organ transplant
5. Receiving other clinical trial medication
6. Already prescribed regular Cayston®

Ages: 16 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Average actual change in percent predicted forced expiratory volume at 1 second (FEV1) from Day 1 to Day 14 | 14 days
  The actual change in FEV1 (%predicted) from Day 1 of admission to Day 7 & Day 14

SECONDARY OUTCOMES:
Time to first pulmonary exacerbation | 12 months
  Time from discharge to next pulmonary exacerbation
Average change from baseline in the Cystic Fibrosis Quality of Life Questionnaire (CFQ-R) | 14 days
  Average change from baseline (Day 1) in the CFQ-R Respiratory Symptom Score (RSS) at the end (Day 14) of each arm of the study
Microbiome changes | 14 days
  Changes in the structure and composition of the microbiome at the beginning and end of each treatment arm
PA sputum counts | 14 days
  Changes in sputum PA counts from the beginning to end of each treatment arm.
Antimicrobial resistance | 14 days
  Prevalence of resistance to antibiotics at the beginning and end of each treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Frost, BMBS BMedSci, Principal Investigator — Liverpool Heart & Chest Hospital NHS Foundation Trust
Locations (1):
- Liverpool Heart & Chest Hospital NHS Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frost F, Young GR, Wright L, Miah N, Smith DL, Winstanley C, Walshaw MJ, Fothergill JL, Nazareth D. The clinical and microbiological utility of inhaled aztreonam lysine for the treatment of acute pulmonary exacerbations of cystic fibrosis: An open-label randomised crossover study (AZTEC-CF). J Cyst Fibros. 2021 Nov;20(6):994-1002. doi: 10.1016/j.jcf.2020.12.012. Epub 2021 Jan 7. PMID 33358119